CLINICAL TRIAL: NCT06433635
Title: Sequential Multiple Assignment Randomized Trial for Bipolar Depression
Acronym: SMART-BD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Dauten Family Center for Bipolar Treatment Innovation, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000831
Record Dates: First submitted 2024-04-22; First posted 2024-05-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bipolar I Disorder; Depression
Keywords: Bipolar; Depression; Adults; Medication
MeSH Terms: conditions — Depression | interventions — cariprazine; Aripiprazole; Escitalopram; Quetiapine Fumarate; Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cariprazine (Experimental)
  Interventions: Drug: Cariprazine
- Aripiprazole /Escitalopram combination (Experimental)
  Interventions: Drug: Aripiprazole/Escitalopram combination
- Quetiapine (Experimental)
  Interventions: Drug: Quetiapine
- Lurasidone (Experimental)
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Cariprazine — 1. Cariprazine monotherapy outperformed placebo in improving depressive symptoms in most large randomized control trials (RCT). Pooled data showed higher remission rates (30.2%) with cariprazine (1.5 mg and 3 mg/day) compared to placebo (20.9%). Its efficacy extends to bipolar I depression, including mixed features and anxiety.
  2. Common adverse effects include nausea (8%) and akathisia (7%). Somnolence and sedation were slightly more common with cariprazine than placebo.
  3. Results from a large RCT evaluating cariprazine for bipolar disorder maintenance treatment (NCT03573297) are awaited. An open-label trial reported reduced manic symptoms over 16 weeks.
  4. Cariprazine is a D3-preferring partial agonist for D3 and D2 receptors. It antagonizes 5-HT2A and 5-HT2B receptors and partially agonizes 5-HT1A receptors. Affinity for 5-HT1C and histamine 1 receptors is low to moderate.
  Other Names: Vraylar
  Arms: Cariprazine
Drug: Aripiprazole/Escitalopram combination — 1. 40-70% of bipolar patients use antidepressants, often with antipsychotics or mood stabilizers. Aripiprazole lacks efficacy in bipolar depression but is used for mania. Escitalopram, studied alongside mood stabilizers, showed some efficacy.
  2. Aripiprazole in bipolar depression trials led to higher rates of akathisia, insomnia, nausea, fatigue, and impulse control disorders. Escitalopram's is generally safe but adverse effects include nausea, diarrhea, insomnia, dry mouth, ejaculatory dysfunction and dizziness.
  3. Aripiprazole monotherapy in bipolar I patients reduced relapse rates and delayed relapse time, but not for depressive episodes.
  4. Aripiprazole acts as a partial agonist at D2, D3, 5-HT1A, and 5-HT2C receptors, with antagonistic effects on α1 and possibly H1 receptors. Escitalopram is highly selective for the serotonin transporter, with no significant activity at other receptors.
  Other Names: Abilify/ Lexapro
  Arms: Aripiprazole /Escitalopram combination
Drug: Quetiapine — 1. Both immediate and extended-release quetiapine monotherapies showed superiority over placebo in acute BD depression across three 8-week randomized trials, confirmed by meta-analysis. Quetiapine exhibited significantly higher remission rates (52.8%) compared to placebo (34.7%) and improved various aspects of life, including quality of life, clinical global impression, sleep, functioning, and anxiety.
  2. Common adverse events of quetiapine include sedation, hypotension, increased appetite, weight gain, dyslipidemia, and elevated glucose levels, particularly in a population already at risk.
  3. Four studies examined quetiapine's maintenance effects in patients with manic, mixed, or depressive episodes. Overall, quetiapine prolonged the time to recurrence for both depressive and manic episodes.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Lurasidone — 1. Lurasidone, either alone or with lithium/valproate, proved more effective than placebo for acute BD depression in two 6-week randomized trials. Remission rates were significantly higher with lurasidone monotherapy (40.9%) and in combination (50.3%) compared to placebo (24.7% and 35.4% respectively). Lurasidone also improved anxiety, quality of life, and disability.
  2. Common mild adverse events included nausea, headache, akathisia, somnolence, sedation, dry mouth, and vomiting. Weight gain, dyslipidemia, and increased glucose levels were not observed.
  3. In a 6-month double-blind discontinuation study post-acute treatment response, lurasidone combined with lithium/valproate prolonged time to depressive episode recurrence compared to placebo (hazard ratio: 0.68). Although not statistically significant due to low placebo recurrence and shorter follow-up, it hints at maintenance efficacy.
  Other Names: Latuda
  Arms: Lurasidone

SUMMARY:
This is a sequential multiple assignment randomized trial for adults (ages > 18) with a bipolar disorder type 1 and type 2 diagnosis currently experiencing a depressive episode. It is a randomized pragmatic trial that will compare four commonly prescribed treatments for bipolar depression, which includes three FDA-approved medications (Cariprazine, Quetiapine and Lurasidone) and one antipsychotic/antidepressant combination (Aripiprazole/Escitalopram).

DETAILED DESCRIPTION:
This is a comparative effectiveness study to address the critical questions of how best to treat people with bipolar disorder who have a major depressive episode: how to get them well, provide second-line treatment when they don't initially get well, and keep them well after they get well. This is a multisite Sequential Multiple Assignment Randomized Trial (SMART) comparative effectiveness design. Investigators will recruit 2726 participants who have BD I or II with a current major depressive episode lasting at least 2 weeks. In Stage 1, investigators will compare four treatment arms, including three FDA approved monotherapies and the most widely used, but understudied, treatment for BD major depressive episode (i.e., a non-FDA approved combination of an antipsychotic and antidepressant). In Stage 2, participants who do not remit will be re-randomized to treatments not used in Stage 1. Investigators will follow all participants for a total of 52 weeks. This study will be conducted in two phases, a feasibility phase and a full study phase. In the feasibility phase, investigators will recruit at 8 of the 19 study sites based on readiness and interest, to ensure the efficacy of the study design before launching the full study phase.

Feasibility Aim 1: To ensure that 8 of the 19 selected sites can recruit, randomize, and retain participants. During the feasibility phase, the selected sites will recruit 133 participants, administer baseline assessments, randomize the participants (at baseline and again at 6-weeks for non-remitters), and conduct follow-up assessments at the end of Stage 1 (6-weeks) and the end of Stage 2 (12-weeks) and end of study (52 weeks or end of feasibility phase, whichever is sooner) and all other scheduled visits.

Feasibility Aim 2: To refine and finalize all study standard operating procedures for the full-scale study. After Aim 1 is complete, any changes in standard operating procedures will be made as needed to be implemented in the full study phase.

Full Scale Study Full-Scale Study Aim 1: To compare the effectiveness, tolerability, and safety of the four treatments for BD major depressive episodes.

Hypothesis 1a: There will be significant differences across the Stage 1 treatments in the proportion of remitters at week 6 (primary endpoint, effectiveness) and in the average adverse event burden and suicidal ideation/behavior at week 6 (secondary endpoints, tolerability and safety).

Hypothesis 1b: Among non-remitters of a given Stage 1 treatment (i.e., participants who do not remit by week 6), there will be significant differences across the three remaining Stage 2 treatments in the proportion of remitters at week 12 (primary endpoint, effectiveness) and the average side effect burden and suicidal ideation/behavior at week 12 (secondary endpoints, tolerability and safety).

Full-Scale Study Aim 2: To characterize the effectiveness, tolerability, and safety of the 12 adaptive interventions for BD major depressive episodes embedded within the SMART design.

Hypothesis 2: On average, there will be significant differences across the 12 embedded adaptive interventions in the proportion of remitters at week 12 (primary endpoint, effectiveness) and in the average side effect burden and suicidal ideation/behavior at week 12 (secondary endpoints, tolerability and safety).

Full-Scale Study Aim 3: To determine individual-level characteristics that predict heterogeneity of treatment effect (HTE) across the 12 adaptive interventions for BD major depressive episodes embedded within the SMART design.

Hypothesis 3a: Individual-level characteristics and symptoms assessed at baseline as well as symptom changes and side effect profiles at week 6 will predict HTE at weeks 12 and 52. Hypothesis 3b: Investigators hypothesize that an optimal personalized adaptive intervention will perform significantly better than the best aggregate embedded adaptive intervention identified in Aim 2 in terms of the proportion of remitters at week 12 (primary endpoint, effectiveness) and the side effect burden and suicidal ideation/behavior at week 12 (secondary endpoints, tolerability and safety).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 years to 75 years
2. Meets criteria for DSM-V Bipolar I or II disorder with a history of manic or hypomanic episodes and current major depressive episode lasting at least 2 weeks
3. Can be managed as an outpatient and participate in the study
4. Willing to be randomized; able to perform study assessments
5. Women of childbearing potential must agree to use adequate contraception (e.g. oral contraceptives, intrauterine device, barrier methods, or total abstinence; Depo Provera is acceptable if it is started 3 months prior to enrollment), and inform staff of their plans to conceive.

Exclusion Criteria:

1. Meets current criteria for a manic episode, rapid cycling within the past year (history of 4 or more mood episodes per year)
2. History of schizophrenia or other nonaffective psychosis
3. Current substance use disorder that will interfere with participation in the study
4. Currently taking the study medications or a history of serious adverse events to any of the study medications, to the extent that as determined by site PI, another trial would not be clinically indicated
5. A history of non-response for depressive episodes, to any of the study medications, when given at adequate doses for at least 6 weeks
6. Current acute suicidal risk that requires inpatient treatment
7. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2726 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
The Remission from Depression Questionnaire | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  RDQ is a 41 items self report questionnaire used to assess the seven domains found in extensive previous research to be important to patients: depressive symptoms, anxiety, coping ability, positive mental health, functioning, life satisfaction and a general sense of well-being. Using a score of 27 as the cutoff, the RDQ scale has a sensitivity of 83.7% and specificity of 77.9% in predicting self-reported remission status. The RDQ has excellent internal consistency reliability (Cronbach's alpha of 0.97 for the total scale and above 0.80 for each of the 7 subscales with test-retest reliability of the total scale = 0.85 and > 0.60 for each subscale). The primary outcome will be remission as defined by a RDQ score < 27. This test will be administered in all assessment visits.
  The RDQ scale ranges from 0-27 per domain, with higher scores indicating greater remission rates.

SECONDARY OUTCOMES:
Safety: Concise Health Risk Tracking Scale | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  CHRT is a 14 item self-report measure of suicidal ideation and behavior in individuals with mood disorders. The CHRT has excellent psychometric properties, with an internal consistency reliability (Cronbach's alpha) of 0.78 and a consistent factor structure with 3 independent factors (current suicidal thoughts and plans, perceived lack of social support, and hopelessness).
  The range is from 14-70, higher scores reflect an increase in suicidality behaviors.
Frequency and Intensity of Side Effects Ratings - Intensity | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  This subscale of the FIBSER scale is a reliable self-report measure of the intensity of side effects from medications in a population receiving treatment for depression. This scale measures the participants side effects intensity from the previous week and has them rate each on a scale from 0-6. The results will help the clinician determine the appropriate level of response.
  The range is from 0-6, higher scores reflect an greater intensity in medication side effects.
Frequency and Intensity of Side Effects Ratings - Frequency | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  This subscale of the FIBSER scale is a reliable and valid self-report measure on the frequency of medication side effects in a population receiving treatment for depression. This scale measures the participants side effects frequency from the previous week and has them rate each on a scale from 0-6. The results will help the clinician determine the appropriate level of response.
  The range is from 0-6, higher scores reflect an greater frequency in medication side effects.
Frequency and Intensity of Side Effects Ratings - Burden | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  This subscale of the FIBSER scale is a reliable self-report measure of the side effects burden of medications in a population receiving treatment for depression. This scale measures the participants side effects burden from the previous week and has them rate each on a scale from 0-6. The results will help the clinician determine the appropriate level of response.
  The range is from 0-6, higher scores reflect an greater burden in medication side effects.

OTHER OUTCOMES:
Altman Self-Rating Mania Scale | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  self-rating mania scale designed to assess the presence and/or severity of manic symptoms in children and adolescents
  The range is from 5-25, higher scores reflect increased symptoms of of mania
Generalized Anxiety Disorder Assessment | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  A seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD).
  The range is from 0-21, higher scores reflect increased symptoms of of anxiety
Medication Reconciliation Tracking Form | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  The MRTF generates the average number of necessary clinical adjustments per month, which provides a method to compare long-term outcomes in a pragmatic trial.
  There is no range or scoring necessary for this assessment.
Patient Health Questionnaire | Investigators will administer this measure every 2 weeks for the first 12 weeks (weeks:0,2,4,6,8,10,12), and then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression
  The range is from 0-27, higher scores reflect increased symptoms of of depression
PROMIS Item Bank v2.0 Cognitive Functioning- Short Form | Investigators will administer this measure at baseline (week 0), week 6, and week 12. Then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  Cognitive deficits will be assessed with the PROMIS- Cognitive Function-Short Form. This 8-item self-report questionnaire has good construct validity and psychometric properties and has been used as an outcome in multiple studies.
  The range is from 8-40, increased scores are associated with a person's increased perception of cognitive function in areas such as concentration, memory, and mental acuity
PROMIS Item Bank v2.0 Satisfaction with Social Roles and Activities | Investigators will administer this measure at baseline (week 0), week 6, and week 12. Then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  This measure is an 8 item self-report questionnaire that assesses the individual's satisfaction with social roles and activities. The measure has clinical validity across a range of chronic conditions, including depression and responds to change in clinical state
  The range is from 8-40 increased scores are associated with higher feelings of satisfaction with performing one's usual social roles and activities
Young Mania Rating Scale | Investigators can administer at any time between weeks 0 to 52. This assessment only applies if patients has a pseudo-remission from depression, indicated if the patient scores a 6 or higher on the self-rated Altman Scale for Rating Mania (ASRM)
  The YMRS is a rating scale used to evaluate manic symptoms at baseline and over time in individuals with mania.
  The range is from 0-60, higher scores reflect increased risk for Bipolar Disorder. If the participant scores 18 or above on the YMRS, they will be considered manic and not in remission even if they meet criteria for remission with the RDQ
Quality of Life Scale | Investigators will administer this measure at baseline (week 0), week 6, and week 12. Then at each study visit during the follow up phase until they are discharged from the study (weeks:20,28,36,44,52 ).
  The QoL.BD93,94 measures 12 core domains (physical, sleep, mood, cognition, leisure, social, spirituality, finances, household, self-esteem, independence, identity) and 2 optional (work, education) domains
  A brief 12-item version represents the core QoL domains and is scored on a five-point range (1: strongly disagree to 5: strongly agree). The range of scoring is 12-60 with higher scores reflecting a greater belief in ones quality of life.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Steve Strakowski, Bloomington, Indiana
  - John Hopkins, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nagy Youssef, Grand Rapids, Michigan
  - University of New Mexico Health Sciences Center Albuquerque, Albuquerque, New Mexico
  - New York University Grossman School of Medicine NYU, New York, New York
  - Montefiore Medical Center and Albert Einstein College of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health Houston Texas, Houston, Texas
- University of British Columbia, Vancouver, British Columbia, Canada